CLINICAL TRIAL: NCT02349321
Title: Skhokho Supporting Success: A Cluster Randomised Controlled Trial of a Multi-faceted, School-based Intimate Partner Violence Primary Prevention Intervention in Gauteng, South Africa
Brief Title: Skhokho Supporting Success: A Cluster RCT of a Multi-faceted, School-based IPV Prevention Intervention in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Research Council, South Africa (Other)
Responsible Party: Principal Investigator, Rachel Jewkes, Professor Rachel K. Jewkes and Dr Anik Gevers, Medical Research Council, South Africa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ECO22-9
Record Dates: First submitted 2015-01-16; First posted 2015-01-28 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Partner of Victim of Physical Abuse
Keywords: physical or sexual intimate partner violence; adolescents; primary prevention; randomised controlled trial; school; South Africa; parenting
MeSH Terms: interventions — Schools

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- School Strengthening (Experimental): Skhokho Supporting Success for Schools: (a) Full year Grade 8 Life Orientation Learner Workbook (following the national curriculum), Educator Guide, and LO Educator support workshops; (b) Educator workshops including values, positive discipline skills, adolescent development, and stress and coping; (c) Learner club workshops (Grade 8s-11s) including creating change for a safe and vibrant school community, human rights at school, communication and conflict resolution skills, and stress and coping.
  Interventions: Behavioral: Skhokho Supporting Success for Schools
- School + Family Strengthening (Experimental): Skhokho Supporting Success for Schools: See description above.
  Skhokho Supporting Success for Families: Participatory four-day workshop for parents/caregivers and their young adolescent children including parallel and joint dialogue sessions. This workshop aims to promote supportive, open relationships between parents/caregivers and their teens and includes communication, negotiation and conflict resolution skills; positive discipline skills; challenging traditional gender constructions; understanding the impact of child abuse; stress and coping.
  Interventions: Behavioral: Skhokho Supporting Success for Schools; Behavioral: Skhokho Supporting Success for Families
- Arm 3: Control (Delayed Intervention) (No Intervention): This group will continue with "treatment as usual" (i.e: school services, activities, and textbooks without specialised intervention). At the end of primary data collection, these schools will be eligible to receive the Schools Strengthening Intervention.

INTERVENTIONS:
Behavioral: Skhokho Supporting Success for Schools — All information describing each facet of the intervention are included in the arm/group descriptions.
  Arms: School + Family Strengthening; School Strengthening
Behavioral: Skhokho Supporting Success for Families — All information describing each facet of the intervention are included in the arm/group descriptions.
  Arms: School + Family Strengthening

SUMMARY:
Development and evaluation of a multi-faceted school-based intervention to prevent intimate partner violence among Grade 8 high school students in South Africa

DETAILED DESCRIPTION:
Primary prevention of intimate partner violence among young men and women requires an intervention which addresses the underlying driving factors of such violence operating at different ecological levels.That is, interventions need to address factors impacting directly on youth and their family relationships, school as an institutional setting. In the school, holistic interventions strengthen the curriculum and teaching, but also the broader environment of learning, including addressing positive discipline and the culture of the school. In order to prevent violence, interventions need to build gender equality, challenge the normative use of violence in schools and homes (e.g., corporal punishment), strengthen teen-adult relationships and communication, and build negotiation and conflict resolution skills, as well as addressing stress and coping.

A three-arm, cluster randomised controlled trial based in high schools in Gauteng, South Africa is evaluating such a multi-faceted primary prevention intervention. This intervention includes school strengthening components for learners and educators, which includes providing a teaching materials for the grade 8 life orientation (LO) curriculum (which covers gender and violence), training teachers in LO teaching, training staff on positive discipline and establishing learner clubs. A second intervention seeks to strengthen families and is a workshop based intervention delivered over 4 day long sessions for a parent or caregiver and their grade 8 adolescent.

The intervention is being evaluated in a three arm randomised controlled trial, with school-level randomisation involving 24 schools. One is a delayed intervention control arm, two arms have the school strengthening intervention and one arm additionally have the family strengthening intervention.

The outcomes will be addressed using qualitative and quantitative methods with data collected from Grade 8 learners (the primary outcome group), school educators and administrators, and parents/caregivers of Grade 8s. These measures will be conducted pre-intervention and at 6, 12, and 18 month follow up periods. In addition, an economic costing evaluation will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* LEARNER/TEEN PARTICIPANTS: enrolled in Grade 8 in one of the study schools; informed consent from parent/guardian to participate in study
* EDUCATOR PARTICIPANTS: currently employed/working as an educator (of any group of learners) at one of the study schools
* PARENT/CAREGIVER PARTICIPANTS: the male or female parent/caregiver/guardian of a Grade 8 learner in Arm 2 schools

Exclusion Criteria:

NONE

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3192 (Estimated)
Dates: Start 2013-02-09 (Actual); Primary Completion 2013-09-30 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
The incidence of IPV (perpetration of physical or sexual IPV for boys and victimisation for girls) | Over 18 months of the study
  Any participant who responds affirmatively to any one of the five questions on physical intimate partner violence or one question on sexual intimate partner violence at the 6, 12 or 18 month data collection points will be deemed to be an incident case of IPV victimisation (if female) or perpetration (if male).
The incidence of severe physical and sexual IPV | Over the last 12 months of the study
  Any participant who responds affirmatively to more than one of the five questions on physical intimate partner violence and/or one question on sexual intimate partner violence at the 12 or 18 month data collection points will be deemed to be an incident case of severe IPV victimisation (if female) or perpetration (if male).

SECONDARY OUTCOMES:
Child-caregiver communication scores | 18 month follow up
  difference in scores derived through summing 5 questions
Childhood trauma scale scores | 18 month follow up
  Difference in scores derived through summing 15 items
The incidence of non-partner rape victimisation and perpetration | Over 18 months of the study
  Any participant who responds affirmatively to any of the non-partner rape questions (2 for girls and 4 for boys) will be deemed to be an incident case of non-partner rape victimisation (if female) and perpetration (if male)
Childhood trauma exposure incidence | 18 month follow up
  Positive affirmation of teens and environment at home Emotional neglect Physical abuse Sexual abuse
Bullying at school score | 18 month follow up
  Comparison of scores across 3 items
Score for communication with girlfriend/boyfriend | 18 month follow up
  Difference in scores measured through summing responses to 5 items
The incidence of emotional Intimate Partner Violence perpetration (for boys) and victimisation (for girls) | 18 months follow up
  Any participant who responds affirmatively to any one of the three questions on emotional intimate partner violence at the 6, 12 or 18 month data collection points will be deemed to be an incident case of emotional IPV victimisation (if female) or perpetration (if male).
the incidence of delinquency | 18-month follow up
  Any participant who responds affirmatively to any one of five questions on delinquency at the 6, 12 or 18 months data collection points will be deemed to be an incident case of delinquency
Depression and anxiety score measured on the Child Depression Inventory | 18-month follow up
  The difference in scores
Gender attitudes score measured across 5 items | 18-month follow up
  the difference in scores

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Jewkes, MD, Principal Investigator — SA Medical Research Council; Anik Gevers, PhD, Principal Investigator — SA Medical Research Council

REFERENCES:
- [Derived] Jewkes R, Gevers A, Chirwa E, Mahlangu P, Shamu S, Shai N, Lombard C. RCT evaluation of Skhokho: A holistic school intervention to prevent gender-based violence among South African Grade 8s. PLoS One. 2019 Oct 29;14(10):e0223562. doi: 10.1371/journal.pone.0223562. eCollection 2019. PMID 31661530
- [Derived] Shamu S, Gevers A, Mahlangu BP, Jama Shai PN, Chirwa ED, Jewkes RK. Prevalence and risk factors for intimate partner violence among Grade 8 learners in urban South Africa: baseline analysis from the Skhokho Supporting Success cluster randomised controlled trial. Int Health. 2016 Jan;8(1):18-26. doi: 10.1093/inthealth/ihv068. Epub 2015 Dec 5. PMID 26637828